CLINICAL TRIAL: NCT01501994
Title: Personalized Approach for Promoting Physical Activity in Mayo Clinic Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Warren G. Thompson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-007103
Record Dates: First submitted 2011-11-29; First posted 2011-12-30 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Weight; Well Being
Keywords: Activity level; Weight; Body Fat; Well Being
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking workstation, counseling, accelerometry feedback (Experimental): 2 week baseline: accelerometer with no feedback 12 experimental: Use of the walking workstation, counseling on increasing activity levels, feedback from the accelerometer 12 week crossover: Feedback from accelerometer, no counseling or walking workstation
  Interventions: Other: GRUVE accelerometer (MUVE, inc.); Other: walking workstation; Procedure: exercise counseling
- Control then crossover (Other): 2 week baseline: accelerometer with no feedback 12 week control period: accelerometer with no feedback 12 week crossover period: accelerometer with feedback, counseling on increasing activity, and use of a walking workstation
  Interventions: Other: GRUVE accelerometer (MUVE, inc.); Other: walking workstation; Procedure: exercise counseling

INTERVENTIONS:
Other: GRUVE accelerometer (MUVE, inc.) — Physicians in the experimental group will be given an accelerometer for 2 weeks (without feedback) prior to starting the study and will continue to have their activity monitored for the duration of the study. The accelerometer monitors movement and accurately estimates physical activity energy expenditure. They will receive feedback about their activity for the remainder of the trial. Physicians in the control group will wear the accelerometer but not receive feedback for the first 14 weeks of the trial. They will receive feedback for the last 12 weeks of the trial as they crossover to the experimental group.
Other: walking workstation — The physicians in the experimental group will be provided with a walking workstation. The walking workstation has a computer keyboard, computer monitor and telephone attached to an exercise treadmill (assembled by the investigators). This allows the user to walk at 1 mile per hour while dictating, typing, responding to e-mail, etc. The treadmill can be placed in an examining room if the physician wishes to use it while dictating notes or it can be placed in a separate office. For the last 12 weeks of the study the experimental group will not use the walking workstation while the control grop will use the workstation (crossover).
  Other Names: treadmill desk
Procedure: exercise counseling — After the first two weeks of baseline data collection, the experimental group will receive exercise counseling for the next 12 weeks. They will be advised to make use of the accelerometer and the walking workstation as well as how to increase their activity in other ways. This group will not receive exercise counseling for the last 12 weeks of the study while the control group will cross over and receive exercise counseling for the last 12 weeks of the study (the control group will not receive exercise counseling for the first 14 weeks of the study).

SUMMARY:
The purpose of the study is to determine if providing physicians with a walking workstation, exercise counseling, and accelerometer feedback about activity will increase physician activity.

DETAILED DESCRIPTION:
20 physicians will be given an activity monitoring accelerometer (GRUVE from MUVE, inc.) for 2 weeks prior to starting the study (without feedback) and will continue to have their activity monitored for the duration of the study. The accelerometer (monitors movement and accurately estimates physical activity energy expenditure). The physicians will be randomized to 12 weeks with accelerometer monitoring but no feedback or counseling (control) or to 12 weeks of accelerometer monitoring (experimental) with feedback about activity levels and 20 minute weekly counseling sessions on how to increase activity (including walking while working). In the 12 week period where physicians receive feedback and counseling, they will also be provided a walking workstation. The walking workstation (assembled by the investigators) has a computer keyboard, computer monitor and telephone attached to an exercise treadmill. This allows the user to walk at 1 mile per hour while dictating, typing, responding to e-mail, etc. The treadmill can be placed in an examining room if the physician wishes to use it while dictating notes or it can be placed in a separate office.

Those physicians assigned to monitoring only for the first 12 weeks will then receive monitoring plus feedback, counseling, and walking workstation use for the next 12 weeks. Those physicians assigned to feedback, counseling, and walking workstation use for the first 12 weeks will continue to receive accelerometer feedback but will no longer receive counseling or use a walking workstation for the subsequent 12 weeks.

Ten physicians will complete the above for the first 26 weeks of the study and 10 physicians will complete the above for the last 26 weeks of the study.

The time line of the study is as follows:

12 Wks Experimental → 12 Wks Control 10 MDs (Wk 1-26) → 2 wks Monitor 12 Wks control → 12 Wks Experimental

12 Wks Experimental → 12 Wks Control 10 MDs (Wk 27-52) → 2 wks Monitor 12 Wks control → 12 Wks Experimental

In summary, physicians use an accelerometer without feedback while in the control group. In the experimental group physicians receive three interventions: accelerometer with feedback, exercise counseling, and the use of a walking workstation (treadmill desk).

ELIGIBILITY:
Inclusion Criteria:

* Physicians working in the Department of Medicine at Mayo Clinic Rochester
* Age 25 to 70 years
* BMI > 25
* Sedentary (exercise for 30 minutes less than 3 times weekly)

Exclusion Criteria:

* Metastatic cancer
* Unable to complete a Bruce protocol exercise stress test
* Planning on retiring in the next 6 months
* Planning on more than 3 weeks of vacation during the 6 month study
* Women of child-bearing age who are pregnant or planning on becoming pregnant.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Activity units determined by accelerometer | 26 weeks

SECONDARY OUTCOMES:
weight in kilograms | 26 weeks
Maximal oxygen consumption (VO2 max) | 26 weeks
  Fitness as determined by an oxygen consumption treadmill test
Percent body fat determined by bone density scan (DEXA) | 26 weeks
Fasting glucose | 26 weeks
Hemoglobin A1c | 26 weeks
Fasting insulin | 26 weeks
Fasting lipid profile | 26 weeks
high sensitivity c-reactive protein | 26 weeks
Well Being using National Center for Health Statistics (NCHS) Well Being Scale | 26 weeks
Depression by Center for Epidemiologic Studies Depression (CES-D) Scale | 26 weeks
Linear Analog Self Assessment Scale | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Warren G Thompson, MD, Principal Investigator — Mayo Clinic